CLINICAL TRIAL: NCT00920387
Title: LSD-assisted Psychotherapy in Persons Suffering From Anxiety Associated With Advanced-stage Life Threatening Diseases. A Phase-II, Double-blind, Placebo-controlled Dose-response Pilot Study
Brief Title: Lysergic Acid Diethylamide (LSD)-Assisted Psychotherapy in People With Illness-related Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LDA1
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Anxiety
Keywords: Anxiety; quality of life; psychotherapy; potentially fatal illness; lysergic acid diethylamide
MeSH Terms: conditions — Anxiety Disorders | interventions — Lysergic Acid Diethylamide; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Dose LSD (200 mcg) (Experimental): 200 mcg LSD administered once during each of two LSD-assisted therapy sessions, scheduled two to four weeks apart.
  Interventions: Drug: 200 mcg LSD; Behavioral: Therapy
- Active Placebo LSD (20 mcg) (Active Comparator): 20 mcg LSD administered once during each of two LSD-assisted therapy sessions, scheduled two to four weeks apart.
  Interventions: Drug: 20 mcg LSD; Behavioral: Therapy

INTERVENTIONS:
Drug: 200 mcg LSD — Administering 200 mcg LSD orally once at the start of each of two day-long psychotherapy session
  Other Names: Lysergic acid diethylamide
  Arms: Full Dose LSD (200 mcg)
Drug: 20 mcg LSD — Administer 20 mcg LSD orally once at the start of each of two day-long psychotherapy session
  Other Names: Lysergic acid diethylamide
  Arms: Active Placebo LSD (20 mcg)
Behavioral: Therapy — Therapy provided by male and female co-therapists

SUMMARY:
This study will find out whether psychotherapy combined with lysergic acid diethylamide (LSD) is safe and is helpful in people who are anxious because they have a potentially fatal disease. The study will measure anxiety and quality of life before and after people have two sessions with either full or active placebo dose of LSD. They expect LSD-assisted psychotherapy to reduce anxiety and improve quality of life.

DETAILED DESCRIPTION:
Diagnosis with a potentially fatal illness is distressing and can provoke anxiety that further reduces quality of life, and a treatment that reduces anxiety when facing deteriorating health and mortality will improve quality of life for people with such illnesses. Forty to fifty years ago, researchers investigated lysergic acid diethylamide (LSD) in combination with psychotherapy to treat anxiety when facing advanced stage cancer. This psychedelic (hallucinogenic) drug can produce transformative or mystical experiences and insights that can help in anxiety reduction. This study will be a randomized, active placebo controlled,double-blind pilot study of the safety and efficacy of LSD-assisted psychotherapy as a way of reducing anxiety in people with potentially fatal illnesses. This study will examine whether two sessions of LSD-assisted psychotherapy scheduled two to four weeks apart will reduce anxiety and improve quality of life for people experiencing anxiety as a result of a potentially fatal illness.

Study subjects will receive either 200 or 20 mcg (micrograms) LSD during two day-long psychotherapy sessions scheduled two to four weeks apart. Subjects in this study will have a 66% of receiving the full dose of 200 mcg LSD, and they have a 33% chance of getting the active placebo dose of 20 mcg LSD. Neither the researchers nor the subject will know whether he got 200 or 20 mcg LSD. Upon participant agreement, all psychotherapy sessions will be recorded to audio and video.

The randomized part of the study will last three and a half months (14 weeks).

People who learn they got the active placebo dose of LSD during the randomized phase can go on to to take part in an "open label" study phase, where they will get the full dose of LSD during two day-long psychotherapy sessions scheduled two to four weeks apart. "Open label" means that they and the researchers will both be aware that they are getting the full dose of LSD.

Participants who received the full dose of LSD and took part in all study visits will be assessed for symptoms of anxiety and depression and quality of life 12 months after their final experimental session.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of advanced-stage potentially fatal illness. As well as metastatic cancer this may include autoimmune, neurological, infectious or rheumatoid diseases as well. The participant must have a probability of survival of more than six months. The estimated life expectancy in relation to the study must be documented.
* The participant makes the decision to participate in the study by his or her own will and that there is no inhibition to his or her will or ability of deciding due to the primary disease.
* Meet DSM-IV criteria for Anxiety Disorder as indicated by the SCID or have a score of at least 40 on each part of the STAI.
* Have failed to respond adequately or at all to medication or psychotherapy intended to reduce anxiety, or have refused to take anxiolytic medication.
* May be diagnosed with another affective disorder other than anxiety disorder, except bipolar-I disorder.
* Are at least 18 years of age.
* Are willing to commit to medication dosing, experimental sessions, follow-up sessions, and to complete evaluation instruments (although they may withdraw from the study at any time without cause).
* Are willing to withdraw from taking any psychiatric medications during the experimental session period. Drugs must be discontinued long enough before the first LSD treatment session to avoid the possibility of a drug-drug interaction (the interval will be at least 5 times the particular drug's half-life).
* If in ongoing psychotherapy, those recruited into the study may continue to see their outside therapist, provided they sign a release for the investigators to communicate directly with their therapist. Participants should not change therapists, increase or decrease the frequency of therapy or commence any new type of therapy until after the evaluation session 2 months after the second LSD treatment session.
* Participants must agree that, for one week preceding each LSD treatment session:
* a. Clinical judgment will be used to determine permissible herbal supplements.
* b. They will not initiate any new prescription medications (except with prior approval of the research team).
* c. Clinical judgment will be used to determine permissible nonprescription medications.
* Participants must be willing to follow restrictions and guidelines concerning consumption of food, beverages and nicotine the night before and just prior to each LSD session.

Exclusion Criteria:

* Women who are pregnant or nursing, or of child bearing potential and are not practicing an effective means of birth control.
* Anyone with past or present diagnosis with a primary psychotic disorder.
* Meeting DSM-IV criteria for Dissociative Disorder or Bipolar-I Affective Disorder.
* Meeting DSM-IV criteria for abuse of or dependence on any substance (other than caffeine or nicotine) in the past 60 days.
* Diagnosed with significant somatic problems, that in the clinical judgment of the investigators poses too great a potential for side effects.
* No sufficient liver function at the baseline examination or the day before the experimental sessions.
* Having evidence of CNS affection from the primary disease (e.g. brain metastasis), shown by neurocognitive impairment.
* Weighing less than 45 kg.
* Reasonably judged to present a serious suicide risk or who are likely to require psychiatric hospitalization during the course of the study.
* Unable to fully understand the potential risks and benefits of the study and give informed consent.
* Requiring ongoing concomitant therapy with a psychotropic drug (other than as needed, anxiety medications, and pain control medications) and are unable or unwilling to comply with the washout period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2011-04-14 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gasser, MD, Principal Investigator — Private practices of Peter Gasser; Swiss Medical Association for Psycholytic Therapy (SAPT)
Locations (1):
- Private Practices of Peter Gasser MD, Solothurn, Switzerland

REFERENCES:
- [Result] Gasser P, Holstein D, Michel Y, Doblin R, Yazar-Klosinski B, Passie T, Brenneisen R. Safety and efficacy of lysergic acid diethylamide-assisted psychotherapy for anxiety associated with life-threatening diseases. J Nerv Ment Dis. 2014 Jul;202(7):513-20. doi: 10.1097/NMD.0000000000000113. PMID 24594678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through general information about the study reported in media, by flyers, presentations in hospitals or cancer support groups, or referral from other physicians.
Groups:
- Full Dose LSD (200 mcg) Blinded Stage 1: 200 mcg LSD administered once during each of two blinded LSD-assisted therapy sessions, scheduled two to four weeks apart during Stage 1
  200 mcg LSD: Administering 200 mcg LSD orally once at the start of each of two day-long psychotherapy session
  Therapy: Therapy provided by male and female co-therapists
- Active Placebo LSD (20 mcg) Stage 1: 20 mcg LSD administered once during each of two blinded LSD-assisted therapy sessions, scheduled two to four weeks apart during Stage 1.
  20 mcg LSD: Administer 20 mcg LSD orally once at the start of each of two day-long psychotherapy session
  Therapy: Therapy provided by male and female co-therapists
- Full Dose LSD (200 mcg) Open-Label Stage 2: 200 mcg LSD administered open-label once during two experimental sessions, scheduled two to eight weeks apart during Stage 2
Period: Stage 1
Arm/Group | Full Dose LSD (200 mcg) Blinded Stage 1 | Active Placebo LSD (20 mcg) Stage 1 | Full Dose LSD (200 mcg) Open-Label Stage 2
Started | 8 | 4 | 0
Completed | 7 | 4 | 0
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Stage 2
Arm/Group | Full Dose LSD (200 mcg) Blinded Stage 1 | Active Placebo LSD (20 mcg) Stage 1 | Full Dose LSD (200 mcg) Open-Label Stage 2
Started | 0 | 0 | 3
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Dose LSD (200 mcg) | Active Placebo LSD (20 mcg) | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (8.4) | 57.4 (9.9) | 51.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
History of suicidal tendencies [Count of Participants; unit: Participants]
  None | 8 | 1 | 9
  Mild | 0 | 2 | 2
Type of life-threatening illness [Count of Participants; unit: Participants]
  Metastatic breast carcinoma | 3 | 1 | 4
  Metastatic gastric carcinoma | 2 | 0 | 2
  Plasmocytoma | 1 | 0 | 1
  Non-Hodgkin's Lymphoma | 0 | 1 | 1
  Celiac Disease | 0 | 1 | 1
  Parkinson's Disease | 1 | 0 | 1
  Bechterew's Disease | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Baseline State-Trait Anxiety Inventory (STAI)
Description: The STAI differentiates between State Anxiety, defined as "anxiety experienced in reaction to a specific environmental circumstance," and Trait Anxiety, defined as "long-standing nervous affect or anxiety disorder." The STAI-state subscale is a 20-item self-reported scale which assesses subjects' levels of transient, situationally oriented, anxiety. Participants respond to each item by selecting a response from a 4-point Likert scale ranging from 4 ("Not at all") to 1 ("Very much so"). STAI-state scores are summed for a total score that range from 20 to 80, with higher scores indicating greater state anxiety. The STAI-trait subscale also consists of 20-items and is scored the same way, with total scores ranging from 20 to 80, with higher scores indicating greater trait anxiety.
Time Frame: Baseline (Visit 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Dose LSD (200 mcg) | Active Placebo LSD (20 mcg)
Number analyzed (Participants) | 8 | 3
score on a scale
  STAI-state | 53.1 (4.7) | 47.7 (7.7)
  STAI-trait | 53.2 (4.3) | 43.3 (7.0)

2. Primary Outcome: Primary Endpoint State-Trait Anxiety Inventory (STAI)
Description: as for outcome 1
Time Frame: 2 months after second experimental session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Dose LSD (200 mcg) | Active Placebo LSD (20 mcg)
Number analyzed (Participants) | 8 | 3
score on a scale
  STAI-state | 41.5 (3.2) | 51.7 (5.3)
  STAI-trait | 45.2 (3.7) | 49.0 (6.1)

ADVERSE EVENTS:
Time Frame: From enrollment to end of Stage 2 (approximately 11 months)
Groups:
- Full Dose LSD (200 mcg Stage 1): 200 mcg LSD administered once during each of two LSD-assisted therapy sessions, scheduled two to four weeks apart.
  200 mcg LSD: Administering 200 mcg LSD orally once at the start of each of two day-long psychotherapy session
  Therapy: Therapy provided by male and female co-therapists
- Active Placebo LSD (20 mcg Stage 1): 20 mcg LSD administered once during each of two LSD-assisted therapy sessions, scheduled two to four weeks apart.
  20 mcg LSD: Administer 20 mcg LSD orally once at the start of each of two day-long psychotherapy session
  Therapy: Therapy provided by male and female co-therapists
- Full Dose LSD (200 mcg Stage 2): 200 mcg LSD administered once during each of two LSD-assisted therapy sessions, scheduled two to eight weeks apart.
  200 mcg LSD: Administering 200 mcg LSD orally once at the start of each of two day-long psychotherapy session
  Therapy: Therapy provided by male and female co-therapists
Arm/Group | Full Dose LSD (200 mcg Stage 1) | Active Placebo LSD (20 mcg Stage 1) | Full Dose LSD (200 mcg Stage 2)
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 8/8 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Dose LSD (200 mcg Stage 1) (N=8) | Active Placebo LSD (20 mcg Stage 1) (N=4) | Full Dose LSD (200 mcg Stage 2) (N=3)
Metastic Esophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pyelonephritis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Full Dose LSD (200 mcg Stage 1) (N=8) | Active Placebo LSD (20 mcg Stage 1) (N=4) | Full Dose LSD (200 mcg Stage 2) (N=3)
Pneumonia (Infections and infestations) | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Palmar-plantar Erythrody Saesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 1
Anger (Psychiatric disorders) | 1 | 2 | 0
Disturbance in Attention (Nervous system disorders) | 0 | 1 | 0
Feeling Cold (General disorders) | 6 | 0 | 1
Affect Liability (Psychiatric disorders) | 1 | 1 | 1
Emotional Distress (Psychiatric disorders) | 5 | 1 | 0
Time Perception Altered (Psychiatric disorders) | 4 | 0 | 2
Thinking Abnormal (Psychiatric disorders) | 1 | 1 | 0
Perseveration (Psychiatric disorders) | 0 | 0 | 1
Tachyphrenia (Psychiatric disorders) | 0 | 1 | 0
Feeling Abnormal (Psychiatric disorders) | 5 | 2 | 1
Derealization (Psychiatric disorders) | 1 | 0 | 1
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Illusions (Psychiatric disorders) | 6 | 1 | 2
Mydriasis (Eye disorders) | 3 | 0 | 0
Perspiration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Impaired Gait (General disorders) | 2 | 0 | 2
Feeling of Relaxation (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Depersonalization (Psychiatric disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Altered Perception of Music (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2010-04-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT00920387/ICF_000.pdf